CLINICAL TRIAL: NCT05335902
Title: The Influence of Extracorporeal Circulation During Cardiac Surgery on Optic Nerve Sheath Diameter
Brief Title: Optic Nerve Sheath After Extracorporeal Circulation
Status: Completed | Type: Observational
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Other Study IDs: UKC-MB-KME-59/21
Record Dates: First submitted 2021-10-29; First posted 2022-04-20 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Disease; Cardiac Valve Disease
Keywords: extracorporeal circulation; otpic nerve sheath diameter; postoperative cognitive disfunction; postoperative nausea and vomiting
MeSH Terms: conditions — Heart Diseases; Heart Valve Diseases; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard cardiopulmonary bypass: patients 18 year or older undergoing heart surgery with standard cardiopulmonary bypass
  Interventions: Diagnostic Test: ultrasound measurement of the optic nerve sheath diameter; Diagnostic Test: MoCA test
- mini-cardiopulmonary bypass: patients 18 year or older undergoing heart surgery with standard mini-cardiopulmonary bypass
  Interventions: Diagnostic Test: ultrasound measurement of the optic nerve sheath diameter; Diagnostic Test: MoCA test

INTERVENTIONS:
Diagnostic Test: ultrasound measurement of the optic nerve sheath diameter — ultrasound measurement of the optic nerve sheath diameter
Diagnostic Test: MoCA test — MoCA test is a short bedside test for measuring cognitive disfunction

SUMMARY:
The purpose of this study is to assess the influence of extracorporeal circulation during cardiac surgery on the optic nerve sheath diameter (ONSD) after the surgery.

DETAILED DESCRIPTION:
ONSD will be measured before and 1 hour after the surgery and in the morning of day 1 after the surgery. Fluid balance and lactate will be measured too. PONV will be assessed. Patients will be evaluated with MoCA test on the day before surgery and on the day 3 after the surgery for cognitive disfunction.

ELIGIBILITY:
Inclusion Criteria:

* heart surgery with use of cardiopulmonary bypass

Exclusion Criteria:

* pregnancy and lactation
* neurologic disorders
* hyperthyroidism
* optic nerve disorders

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older which are scheduled for heart surgery (coronary bypass, valve disease, thoracic aortic disease) in which cardiopulmonary bypass is used.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound measuring of optic nerve sheath diameter baseline | Before start of surgery
  Baseline optic nerve sheath diameter measurement before start of surgery with a linear ultrasound probe (Scan) in coronal and axial plane
Ultrasound measuring of optic nerve sheath diameter end of surgery | 1 hour after the end of surgery
  Optic nerve sheath diameter measurement 1 hour after the end of surgery with a linear ultrasound probe in coronal and axial plane
Ultrasound measuring of optic nerve sheath diameter day 1 | day 1 after the surgery
  Optic nerve sheath diameter measurement in the morning on day 1 after the surgery with a linear ultrasound probe in coronal and axial plane

SECONDARY OUTCOMES:
postoperative cognitive disfunction measured with the MoCA test | on the day before surgery, on day 3 after the surgery
  MoCA test is a validated test for cognitive disfunction, especially in patients who are elderly than 60 years, the study is comparing the MoCA test values on the day before surgery with the values on day 3 after the surgery
postoperative nausea and vomiting (PONV) | during the first 24 hours after surgery
  Postoperative nausea and vomiting is common after cardiac surgery, the occurrence of postoperative nausea and vomiting will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- University medical centre Maribor, Maribor, Slovenia

REFERENCES:
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Selnes OA, Goldsborough MA, Borowicz LM, McKhann GM. Neurobehavioural sequelae of cardiopulmonary bypass. Lancet. 1999 May 8;353(9164):1601-6. doi: 10.1016/S0140-6736(98)07576-X. PMID 10334272
- [Background] Zamvar V, Williams D, Hall J, Payne N, Cann C, Young K, Karthikeyan S, Dunne J. Assessment of neurocognitive impairment after off-pump and on-pump techniques for coronary artery bypass graft surgery: prospective randomised controlled trial. BMJ. 2002 Nov 30;325(7375):1268. doi: 10.1136/bmj.325.7375.1268. PMID 12458242
- [Background] Bayram H, Hidiroglu M, Cetin L, Kucuker A, Iriz E, Uguz E, Saglam F, Sener E. Comparing S-100 beta protein levels and neurocognitive functions between patients undergoing on-pump and off-pump coronary artery bypass grafting. J Surg Res. 2013 Jun 15;182(2):198-202. doi: 10.1016/j.jss.2012.10.047. Epub 2012 Nov 9. PMID 23183054
- [Background] Stroobant N, Van Nooten G, Belleghem Y, Vingerhoets G. Short-term and long-term neurocognitive outcome in on-pump versus off-pump CABG. Eur J Cardiothorac Surg. 2002 Oct;22(4):559-64. doi: 10.1016/s1010-7940(02)00409-8. PMID 12297172
- [Background] Riha H, Drabek T, Polisenska J, Brezina A. Postoperative nausea and vomiting in cardiac surgery. Eur J Anaesthesiol. 2009 Jun;26(6):535-6. doi: 10.1097/eja.0b013e328320a67a. No abstract available. PMID 19445063
- [Background] Gong Z, Li J, Zhong Y, Guan X, Huang A, Ma L. Effects of dexmedetomidine on postoperative cognitive function in patients undergoing coronary artery bypass grafting. Exp Ther Med. 2018 Dec;16(6):4685-4689. doi: 10.3892/etm.2018.6778. Epub 2018 Sep 19. PMID 30542420
- [Background] Styra R, Larsen E, Dimas MA, Baston D, Elgie-Watson J, Flockhart L, Lindsay TF. The effect of preoperative cognitive impairment and type of vascular surgery procedure on postoperative delirium with associated cost implications. J Vasc Surg. 2019 Jan;69(1):201-209. doi: 10.1016/j.jvs.2018.05.001. Epub 2018 Jun 22. PMID 29941317
- [Background] O'Dwyer C, Prough DS, Johnston WE. Determinants of cerebral perfusion during cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 1996 Jan;10(1):54-64; quiz 65. doi: 10.1016/s1053-0770(96)80179-0. PMID 8634388
- [Background] Barbosa Nde F, Cardinelli DM, Ercole FF. Determinants of neurological complications with the use of extracorporeal circulation (ECC). Arq Bras Cardiol. 2010 Dec;95(6):e151-7. doi: 10.1590/s0066-782x2010001600022. No abstract available. English, Portuguese, Spanish. PMID 21271187
- [Background] Salameh A, Dhein S, Dahnert I, Klein N. Neuroprotective Strategies during Cardiac Surgery with Cardiopulmonary Bypass. Int J Mol Sci. 2016 Nov 21;17(11):1945. doi: 10.3390/ijms17111945. PMID 27879647
- [Background] Murphy GJ, Angelini GD. Side effects of cardiopulmonary bypass: what is the reality? J Card Surg. 2004 Nov-Dec;19(6):481-8. doi: 10.1111/j.0886-0440.2004.04101.x. PMID 15548178
- [Background] Hirleman E, Larson DF. Cardiopulmonary bypass and edema: physiology and pathophysiology. Perfusion. 2008 Nov;23(6):311-22. doi: 10.1177/0267659109105079. PMID 19454559
- [Background] Ottens TH, Hendrikse J, Slooter AJ, van Herwerden LA, Dieleman JM, van Dijk D. Low incidence of early postoperative cerebral edema after coronary artery bypass grafting. J Cardiothorac Vasc Anesth. 2015;29(3):632-6. doi: 10.1053/j.jvca.2014.12.004. Epub 2014 Dec 3. PMID 25817849
- [Background] Harris DN, Oatridge A, Dob D, Smith PL, Taylor KM, Bydder GM. Cerebral swelling after normothermic cardiopulmonary bypass. Anesthesiology. 1998 Feb;88(2):340-5. doi: 10.1097/00000542-199802000-00011. PMID 9477053
- [Background] Harris DN, Bailey SM, Smith PL, Taylor KM, Oatridge A, Bydder GM. Brain swelling in first hour after coronary artery bypass surgery. Lancet. 1993 Sep 4;342(8871):586-7. doi: 10.1016/0140-6736(93)91412-f. PMID 8102722
- [Background] Linardi D, Walpoth B, Mani R, Murari A, Tessari M, Hoxha S, Anderloni M, Decimo I, Dolci S, Nicolato E, Bontempi P, Merigo F, Luciani GB, Faggian G, Rungatscher A. Slow versus fast rewarming after hypothermic circulatory arrest: effects on neuroinflammation and cerebral oedema. Eur J Cardiothorac Surg. 2020 Oct 1;58(4):792-800. doi: 10.1093/ejcts/ezaa143. PMID 32408343
- [Background] Cheung AT, Messe SR. Preventing Brain Injury After Cardiopulmonary Bypass Will Require More Than Just Dialing Up the Pressure. Circulation. 2018 Apr 24;137(17):1781-1783. doi: 10.1161/CIRCULATIONAHA.118.033197. No abstract available. PMID 29685929
- [Background] Evensen KB, Eide PK. Measuring intracranial pressure by invasive, less invasive or non-invasive means: limitations and avenues for improvement. Fluids Barriers CNS. 2020 May 6;17(1):34. doi: 10.1186/s12987-020-00195-3. PMID 32375853
- [Background] Chen H, Ding GS, Zhao YC, Yu RG, Zhou JX. Ultrasound measurement of optic nerve diameter and optic nerve sheath diameter in healthy Chinese adults. BMC Neurol. 2015 Jul 7;15:106. doi: 10.1186/s12883-015-0361-x. PMID 26148482
- [Background] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900
- [Background] Aduayi OS, Asaleye CM, Adetiloye VA, Komolafe EO, Aduayi VA. Optic nerve sonography: A noninvasive means of detecting raised intracranial pressure in a resource-limited setting. J Neurosci Rural Pract. 2015 Oct-Dec;6(4):563-7. doi: 10.4103/0976-3147.165347. PMID 26752428
- [Background] Tawfik EA, Walker FO, Cartwright MS. Neuromuscular ultrasound of cranial nerves. J Clin Neurol. 2015 Apr;11(2):109-21. doi: 10.3988/jcn.2015.11.2.109. PMID 25851889
- [Background] Ali MA, Hashmi M, Shamim S, Salam B, Siraj S, Salim B. Correlation of Optic Nerve Sheath Diameter with Direct Measurement of Intracranial Pressure through an External Ventricular Drain. Cureus. 2019 Sep 26;11(9):e5777. doi: 10.7759/cureus.5777. PMID 31723536
- [Background] Yilmaz G, Akca A, Kiyak H, Salihoglu Z. Elevation in optic nerve sheath diameter due to the pneumoperitoneum and Trendelenburg is associated to postoperative nausea, vomiting and headache in patients undergoing laparoscopic hysterectomy. Minerva Anestesiol. 2020 Mar;86(3):270-276. doi: 10.23736/S0375-9393.19.13920-X. Epub 2019 Oct 28. PMID 31680498
- [Background] Hu J, Li CJ, Wang BJ, Li XY, Mu DL, Wang DX. The sensitivity and specificity of statistical rules for diagnosing delayed neurocognitive recovery with Montreal cognitive assessment in elderly surgical patients: A cohort study. Medicine (Baltimore). 2020 Jul 17;99(29):e21193. doi: 10.1097/MD.0000000000021193. PMID 32702882